CLINICAL TRIAL: NCT02431000
Title: Male Fertility Pre- and Post- Radiation and Chemotherapy, and Sperm Preservation
Brief Title: Male Fertility and Sperm Cryopreservation
Status: Withdrawn | Type: Observational
Why Stopped: PI is no longer at this University.
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: 12-02277-XP
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2019-01

CONDITIONS: Fertility; SPERM; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Sperm Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subject who express the desire to have pre-treatment sperm cryopreservation. These subjects will undergo an informed consent process. If the five years of storage are up before subjects are ready to claim it, it will be their responsibility to keep the account open by paying a fee of about $300.00 per any additional year in storage. If they withdraw from the study before the five years are up, they will be free to claim the sperm from storage or to leave it there until the five years are up. Afterwards, they will be responsible for the annual fees.
  Long term Semen Freezing :
  After freezing, sperm samples will be sent to FairFax Cryobank in Austin, Texas for long-term storage. A storage agreement plan has been pre-arranged with FairFax and UTMG.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Male Chemo/Radiotherapy Candidates: Adult and post-pubertal males, 13 years of age or older, presenting to clinic because diagnosed with cancer, who wish to preserve their future fertility. Sperm and blood collected for analysis. If minors, parents or guardians have to give consent to the procedure while the boys give their assent.
  This is a prospective observational cohort study.
  Interventions: Procedure: Sperm and blood collected for analysis

INTERVENTIONS:
Procedure: Sperm and blood collected for analysis — Sperm Collection and Freezing (Cryopreservation), Blood Collection for analysis

SUMMARY:
PURPOSE: Primary objective: To assess the feasibility and outcomes of male fertility preservation by sperm freezing prior to starting treatment requiring alkylating agents and/or total body irradiation.

Secondary objective: To assess pre- and post-treatment sperm production and hormonal status by measurement of serum anti-mullerian hormone (AMH), inhibin-B, follicle stimulating hormone (FSH), luteinizing hormone (LH), testosterone, and androstendione.

DETAILED DESCRIPTION:
RATIONALE: In June 2006, the American Society of Clinical Oncology published a series of recommendations on fertility preservation for patients with cancer, concluding that "To preserve the full range of options, fertility preservation, approaches should be considered as early as possible during treatment planning". These guidelines reflect the greater attention that has been given in recent years to the fertility complications that can occur as a result of cancer treatment (eg, chemotherapies and radiation).

Different cancer treatments such as cytotoxic therapy can lead to azoospermia and sterility for an unknown period. Whether the type of cancer significantly affects semen quality or not is under debate. In some studies, semen quality of cancer patients did not differ significantly from those without, but other studies have indicated a significant decrease in sperm quality in some malignancies such as testicular cancer and Hodgkin. Fertility and reproductive function are the principal concerns in 80% of successfully treated men with cancer. Although cancer survivors can become parents by adoption or gamete donation, most would prefer to have biologic parenthood and biologically related children.

POPULATION: Adult and post-pubertal males, 13 years of age or older, presenting to our clinic because diagnosed with cancer, who wish to preserve their future fertility. If minors, parents or guardians have to give consent to the procedure while the boys give their assent.

DESIGN: This is a prospective observational cohort study.

PROCEDURES: Subject Recruitment and Screening Subjects will be recruited by referral from the Memphis area cancer centers and physicians whose patients express the desire to have pre-treatment sperm cryopreservation. Minors will be recruited by referral from the St. Jude Children's Research Hospital (SJCRH) and Methodist-Le Bonheur physicians. These subjects will undergo an informed consent process in accordance with University of Tennessee Health Science Center and SJCRH Institutional Review Board. If the five years of storage are up before subjects are ready to claim it, it will be their responsibility to keep the account open by paying a fee of about $300.00 per any additional year in storage. If they withdraw from the study before the five years are up, they will be free to claim the sperm from storage or to leave it there until the five years are up. Afterwards, they will be responsible for the annual fees.

Long term Semen Freezing :

After freezing, sperm samples will be sent to FairFax Cryobank in Austin, Texas for long-term storage. A storage agreement plan has been pre-arranged with FairFax and University of Tennessee Medical Group.

Follow-up clinical information will be collected only when patients return for fertility treatment, if coming to our facility.

No follow-up evaluation will be performed if the patients decide to have their specimens shipped to their new hometown or fertility clinic. However, patients will be asked to contact the investigators regarding their serum/tissue sample use and fertility outcomes. If no contact in this regard is made, patients will be re-contacted by the investigators once every year, if at that time they are 18 years old, or older, and if the five-year storage has expired.

ELIGIBILITY:
Inclusion Criteria:

* male, aged 13 years or older,
* diagnosed with cancer, but not yet undergoing therapy
* willing to participate in this clinical trial
* signed Informed consent document

Exclusion Criteria:

* under 13 years old
* have already begun Chemo or radiotherapy

Min Age: 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject Recruitment and Screening Subjects will be recruited by referral from the Memphis area cancer centers and physicians whose patients express the desire to have pre-treatment sperm cryopreservation. Minors will be recruited by referral from the SJCRH and Methodist-Le Bonheur physicians
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Semen and lab parameters pre-cancer treatment. | On Day 1/Visit 1 (1 hour and 30 minutes)
  •Semen Collection during an office visit. If no sample is able to be collected at that time, the visit may be rescheduled for another day. Also, 2 tablespoons of blood will be drawn from the arm by needle stick for hormonal blood tests. Information such as age, weight, and height, and medical history such as previous health problems will be copied from the medical record.
Semen and lab parameters post-cancer treatment. | Day 2/ Visit 2; 4 months after the completion of chemotherapy or radiotherapy
  Semen Collection during an office visit. If no sample is able to be collected at that time, the visit may be rescheduled for another day. Also, 2 tablespoons of blood will be drawn from the arm by needle stick for hormonal blood tests. Information such as age, weight, and height, and medical history such as previous health problems will be copied from the medical record.

SECONDARY OUTCOMES:
Pre-therapy thawing evaluation of specific biochemical markers in the serum and in semen samples. | On average,analysis will occur within 6 months of the completion of the subject's participation.
  Semen will be frozen following existing freezing protocols. Fifty microliters (50 mL), each specimen, will be stored in formalin for later immunohistochemical examination. Fifty mLs will be frozen for metabolite, protein, and messenger Ribonucleic Acid (mRNA) analyses. These analyses will allow us to understand which sperm function is altered by cancer treatment and possibly identify protective measures to prevent such damage. Analyses will be conducted for all samples in the laboratory of the University of Tennessee Center for Reproductive Medicine at the University of Tennessee Health Science Center. This will allow us to have the same reference ranges for each of the different parameters measured and have a homogeneous evaluation of the results. The sperm specimens will be kept in the laboratory until analyzed and/or until completion of the research study.
  Serum hormones levels of all samples from thawed serum samples will be analyzed in a central laboratory (LabCorp).
Post-therapy thawing evaluation of specific biochemical markers in the serum and in semen samples. | On average,analysis will occur within 6 months of the completion of the subject's participation.
  Semen will be frozen following existing freezing protocols. Fifty mLs of each specimen will be stored in formalin for later immunohistochemical examination. Another 50 mLs will be frozen for metabolite, protein, and messenger Ribo Nucleic Acid analyses. These analyses will allow us to understand which sperm function is altered by cancer treatment and possibly identify protective measures to prevent such damage. Analyses will be conducted for all samples in the laboratory of the University of Tennessee Center for Reproductive Medicine at the University of Tennessee Health Science Center. This will allow us to have the same reference ranges for each of the different parameters measured and have a homogeneous evaluation of the results. The sperm specimens will be kept in the laboratory until analyzed and/or until completion of the research study.
  Serum levels of the various hormones will be evaluated for all samples from thawed serum samples in a central laboratory (LabCorp).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Detti, M.D., Principal Investigator — Associate Professor, UTennessee Health Science Center
Locations (1):
- University of Tennessee Health Science Center Center for Reproductive Medicine, ROH,, Memphis, Tennessee, United States

REFERENCES:
- [Result] Bahadur G. Fertility issues for cancer patients. Mol Cell Endocrinol. 2000 Nov 27;169(1-2):117-22. doi: 10.1016/s0303-7207(00)00364-6. PMID 11155943
- [Result] Lee SJ, Schover LR, Partridge AH, Patrizio P, Wallace WH, Hagerty K, Beck LN, Brennan LV, Oktay K; American Society of Clinical Oncology. American Society of Clinical Oncology recommendations on fertility preservation in cancer patients. J Clin Oncol. 2006 Jun 20;24(18):2917-31. doi: 10.1200/JCO.2006.06.5888. Epub 2006 May 1. PMID 16651642
- [Result] Lass A, Akagbosu F, Abusheikha N, Hassouneh M, Blayney M, Avery S, Brinsden P. A programme of semen cryopreservation for patients with malignant disease in a tertiary infertility centre: lessons from 8 years' experience. Hum Reprod. 1998 Nov;13(11):3256-61. doi: 10.1093/humrep/13.11.3256. PMID 9853891
- [Result] Rofeim O, Gilbert BR. Normal semen parameters in cancer patients presenting for cryopreservation before gonadotoxic therapy. Fertil Steril. 2004 Aug;82(2):505-6. doi: 10.1016/j.fertnstert.2003.12.045. PMID 15302317
- [Result] Puscheck E, Philip PA, Jeyendran RS. Male fertility preservation and cancer treatment. Cancer Treat Rev. 2004 Apr;30(2):173-80. doi: 10.1016/j.ctrv.2003.07.005. PMID 15023435
- [Result] Sabanegh ES Jr, Ragheb AM. Male fertility after cancer. Urology. 2009 Feb;73(2):225-31. doi: 10.1016/j.urology.2008.08.474. Epub 2008 Nov 26. PMID 19036419
- [Result] Schover LR. Rates of postcancer parenthood. J Clin Oncol. 2009 Jan 20;27(3):321-2. doi: 10.1200/JCO.2008.19.7749. Epub 2008 Dec 15. No abstract available. PMID 19075256
- [Result] Skinner R, Wallace WH, Levitt GA; UK Children's Cancer Study Group Late Effects Group. Long-term follow-up of people who have survived cancer during childhood. Lancet Oncol. 2006 Jun;7(6):489-98. doi: 10.1016/S1470-2045(06)70724-0. PMID 16750499
- [Result] Williams DH 4th, Karpman E, Sander JC, Spiess PE, Pisters LL, Lipshultz LI. Pretreatment semen parameters in men with cancer. J Urol. 2009 Feb;181(2):736-40. doi: 10.1016/j.juro.2008.10.023. Epub 2008 Dec 16. PMID 19091343